CLINICAL TRIAL: NCT04485546
Title: An 8-week, Multicenter, Open Label, Prospective Study With 24 Weeks of Follow-up to Evaluate Safety and Efficacy of OXERVATE® 0.002% (20 mcg/mL) Cenegermin-bkbj Ophthalmic Solution in Patients With Stage 1 Neurotrophic Keratitis (NK)
Brief Title: Study to Evaluate OXERVATE® in Patients With Stage 1 Neurotrophic Keratitis
Acronym: DEFENDO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dompé Farmaceutici S.p.A (Industry)
Collaborators: Dompé US (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NGF0120
Record Dates: First submitted 2020-07-21; First posted 2020-07-24 (Actual); Results first posted 2023-06-23 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Neurotrophic Keratitis
Keywords: Stage 1 Neurotrophic Keratitis; Corneal Disease; Ocular Disease
MeSH Terms: conditions — Corneal Diseases | interventions — cenegermin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- OXERVATE® 0.002% (20 mcg/mL) cenegermin-bkbj (Experimental): cenegermin-bkbj ophtalmic solution administered as one drop in affected eye(s) every 2 hours 6 times daily for 8 weeks
  Interventions: Drug: cenegermin-bkbj

INTERVENTIONS:
Drug: cenegermin-bkbj — OXERVATE® 0.002% (20 mcg/mL) cenegermin-bkbj ophthalmic solution administered as one drop in the affected eye(s), 6 times a day at 2-hour intervals for 8 weeks, in patients with Stage 1 neurotrophic keratitis.
  Other Names: OXERVATE® 0.002% (20 mcg/mL) cenegermin-bkbj ophthalmic solution

SUMMARY:
This study is to evaluate the safety and efficacy of OXERVATE® 0.002% (20 mcg/mL) cenegermin-bkbj ophthalmic solution in patients with Stage 1 neurotrophic keratitis (NK).

DETAILED DESCRIPTION:
This is a 8-week, multicenter, open label, prospective study with 24 weeks of follow-up to evaluate safety and efficacy of OXERVATE® 0.002% (20 mcg/mL) cenegermin-bkbj ophthalmic solution in patients with Stage 1 neurotrophic keratitis (NK)

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged ≥ 18 years.
2. Patients with Stage 1 NK defined by the Mackie criteria

Exclusion Criteria:

1. Evidence of an active ocular infection (bacterial, viral, protozoal) in either eye.
2. Have current or history of conditions that may confound the study data including but not limited to Ocular Cicatricial Pemphigoid (OCP), Graft Versus Host Disease (GVHD), neuromyelitis optica, uncontrolled dry eye, and Steven Johnson's syndrome.
3. History of severe systemic allergy or severe ocular allergy (including seasonal conjunctivitis expected during the subject's participation in the trial) or chronic conjunctivitis and/or keratitis other than dry eye disease.
4. Patients with severe vision loss with no potential for visual improvement in the study eye, in the opinion of the investigator, or if the subject is deemed legally blind.
5. Ocular surgery or elective ocular surgery expected during participation in the trial.
6. Patients with eyelid abnormality that may alter eyelid function including but not limited to Blepharospasm, Cerebrovascular accident, entropion, ectropion, floppy lid syndrome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2020-09-09 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2022-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Flavio Mantelli, MD, PhD, Study Chair — Domp Farmaceutici SpA
Locations (5):
- United States (5):
  - San Diego, San Diego, California
  - Edgewood, Edgewood, Kentucky
  - Boston, Boston, Massachusetts
  - Saint Louis, St Louis, Missouri
  - Philadelphia, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mastropasqua L, Massaro-Giordano G, Nubile M, Sacchetti M. Understanding the Pathogenesis of Neurotrophic Keratitis: The Role of Corneal Nerves. J Cell Physiol. 2017 Apr;232(4):717-724. doi: 10.1002/jcp.25623. Epub 2016 Oct 17. PMID 27683068
- [Derived] Hamrah P, Massaro-Giordano M, Schanzlin D, Holland E, Berdy G, Goisis G, Pasedis G, Mantelli F. Phase IV Multicenter, Prospective, Open-Label Clinical Trial of Cenegermin (rhNGF) for Stage 1 Neurotrophic Keratopathy (DEFENDO). Ophthalmol Ther. 2024 Feb;13(2):553-570. doi: 10.1007/s40123-023-00866-y. Epub 2024 Jan 4. PMID 38175466

RESULTS

PARTICIPANT FLOW:
Groups:
- OXERVATE® 0.002% (20 mcg/mL) Cenegermin-bkbj: cenegermin-bkbj: Cenegermin-bkbj ophthalmic solution administered as one drop in affected eye(s) every 2 hours 6 times daily for 8 weeks
Period: Overall Study
Arm/Group | OXERVATE® 0.002% (20 mcg/mL) Cenegermin-bkbj
Started | 37
Completed | 29
Not Completed | 8

BASELINE CHARACTERISTICS:
Arm/Group | OXERVATE® 0.002% (20 mcg/mL) Cenegermin-bkbj
Number analyzed (Participants) | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.6 (11.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 35
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 32
  Race: Black or African American | 3
  Race: Asian | 1
  Race: Other | 1
Region of Enrollment [Number; unit: participants]
  United States | 37
Treated Eyes [Number; unit: participants]
  Participants with Treated Study Eye | 37
  Participants with Treated Non-Study Eye | 15

OUTCOME MEASURES:

1. Primary Outcome: Corneal Epithelial Healing
Description: Percentage of patients who experienced corneal epithelial healing. Corneal epithelial healing was defined by the central reading center as the absence of persistent epithelial staining abnormalities related to disease.
Time Frame: Week 8
Population: Full Analysis Set (FAS) - All enrolled patients who received at least one dose of the study drug. The FAS was used both for efficacy and safety analyses. Observed cases (n=33)
Measure: Count of Participants; unit: Participants
Arm/Group | OXERVATE® 0.002% (20 mcg/mL) Cenegermin-bkbj
Number analyzed (Participants) | 33
Participants
  No | 5
  Yes | 28

ADVERSE EVENTS:
Time Frame: 34 Weeks
Description: An AE was defined as any untoward medical occurrence in a patient or clinical investigation patient administered a pharmaceutical product that did not necessarily have a causal relationship with this treatment.
  Safety evaluations were based on adverse event (AE) monitoring, intraocular pressure (IOP), slit lamp exam, and external eye exam.
Groups:
- OXERVATE® 0.002% (20 mcg/mL) Cenegermin-bkbj - Study Eye: cenegermin-bkbj: Cenegermin-bkbj ophthalmic solution administered as one drop in affected eye(s) every 2 hours 6 times daily for 8 weeks - Study Eye
- OXERVATE® 0.002% (20 mcg/mL) Cenegermin-bkbj - Non Study Eye: cenegermin-bkbj: Cenegermin-bkbj ophthalmic solution administered as one drop in affected eye(s) every 2 hours 6 times daily for 8 weeks - Non Study Eye
- OXERVATE® 0.002% (20 mcg/mL) Cenegermin-bkbj - Systemic: enegermin-bkbj: Cenegermin-bkbj ophthalmic solution administered as one drop in affected eye(s) every 2 hours 6 times daily for 8 weeks - Systemic Conditions
Arm/Group | OXERVATE® 0.002% (20 mcg/mL) Cenegermin-bkbj - Study Eye | OXERVATE® 0.002% (20 mcg/mL) Cenegermin-bkbj - Non Study Eye | OXERVATE® 0.002% (20 mcg/mL) Cenegermin-bkbj - Systemic
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/37 | 1/37
Serious Adverse Events (participants affected / at risk) | 1/37 | 0/37 | 7/37
Other Adverse Events (participants affected / at risk) | 22/37 | 13/37 | 16/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OXERVATE® 0.002% (20 mcg/mL) Cenegermin-bkbj - Study Eye (N=37) | OXERVATE® 0.002% (20 mcg/mL) Cenegermin-bkbj - Non Study Eye (N=37) | OXERVATE® 0.002% (20 mcg/mL) Cenegermin-bkbj - Systemic (N=37)
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1
COVID-19 (Infections and infestations) | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 1
Hiatus Hernia (Gastrointestinal disorders) | 0 | 0 | 1
Incarcerated parastomal hernia (Injury, poisoning and procedural complications) | 0 | 0 | 1
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 1
Deep Vein Thrombosis (Vascular disorders) | 0 | 0 | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Iridocyclitis (Eye disorders) | 1 | 0 | 0
Intestinal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
COVID-19 Pneumonia (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OXERVATE® 0.002% (20 mcg/mL) Cenegermin-bkbj - Study Eye (N=37) | OXERVATE® 0.002% (20 mcg/mL) Cenegermin-bkbj - Non Study Eye (N=37) | OXERVATE® 0.002% (20 mcg/mL) Cenegermin-bkbj - Systemic (N=37)
Corneal Dystrophy (Congenital, familial and genetic disorders) | 2 | 1 | 0 — 2 Participants - 1 Case is OU (oculus uterque)
Thyroid Mass (Endocrine disorders) | 0 | 0 | 1
Blepharospasm (Eye disorders) | 1 | 1 | 0 — 1 Participant - Case is OU (oculus uterque)
Conjunctival hyperaemia (Eye disorders) | 2 | 1 | 0 — 2 Participants - 1 Case is OU (oculus uterque)
Contact lens intolerance (Eye disorders) | 0 | 1 | 0
Corneal Oedema (Eye disorders) | 2 | 1 | 0
Diplopia (Eye disorders) | 1 | 1 | 0 — 1 Participant - Case is OU (oculus uterque)
Dry Eye (Eye disorders) | 4 | 2 | 0 — 4 Participants - 2 Cases are OU (oculus uterque)
Ectropion (Eye disorders) | 0 | 1 | 0
Eye irritation (Eye disorders) | 3 | 2 | 0 — 3 Participants - 2 Cases are OU (oculus uterque)
Eye Pain (Eye disorders) | 14 | 2 | 0 — 14 Participants - 2 Cases are OU (oculus uterque)
Eyelid disorder (Eye disorders) | 1 | 0 | 0
Eyelid irritation (Eye disorders) | 1 | 1 | 0 — 1 Participant - Case is OU (oculus uterque)
Eyelid margin crusting (Eye disorders) | 1 | 1 | 0 — 1 Participant - Case is OU (oculus uterque)
Eyelid pain (Eye disorders) | 3 | 2 | 0 — 3 Participants - 2 Cases are OU (oculus uterque)
Foreign body sensation in eyes (Eye disorders) | 4 | 0 | 0
Keratitis (Eye disorders) | 2 | 1 | 0 — 2 Participants - 1 Case is OU (oculus uterque)
Neurotrophic keratopathy (Eye disorders) | 1 | 1 | 0 — 1 Participant - Case is OU (oculus uterque)
Ocular hyperaemia (Eye disorders) | 1 | 0 | 0
Periorbital pain (Eye disorders) | 1 | 0 | 0
Photophobia (Eye disorders) | 1 | 0 | 0
Vision blurred (Eye disorders) | 7 | 3 | 0 — 7 Participants - 3 Cases are OU (oculus uterque)
Visual acuity reduced (Eye disorders) | 1 | 0 | 0
Visual impairment (Eye disorders) | 1 | 1 | 0 — 1 Participant - Case is OU (oculus uterque)
Vitreous Floaters (Eye disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 1
Facial pain (General disorders) | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 1
Secretion discharge (General disorders) | 2 | 1 | 0 — 2 Participants - 1 Case is OU (oculus uterque)
Swelling face (General disorders) | 0 | 0 | 1
Graft versus host disease (Immune system disorders) | 0 | 0 | 1
Conjunctivitis bacterial (Infections and infestations) | 1 | 1 | 0 — 1 Participant - Case is OU (oculus uterque)
Herpes ophthalmic (Infections and infestations) | 1 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 1 | 0
Ophthalmic herpes simplex (Infections and infestations) | 2 | 0 | 0
Ophthalmic herpes zoster (Infections and infestations) | 1 | 0 | 0
Persistent corneal epithelial defect (Injury, poisoning and procedural complications) | 1 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Tooth injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Ocular hypertension (Eye disorders) | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Apraxia (Nervous system disorders) | 1 | 0 | 0
Burning sensation (Nervous system disorders) | 3 | 1 | 0 — 3 Participants - 1 Case is OU (oculus uterque)
Headache (Nervous system disorders) | 0 | 0 | 2
Migraine (Nervous system disorders) | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1
Breast dysplasia (Reproductive system and breast disorders) | 0 | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 1
Subgaleal haematoma (Vascular disorders) | 0 | 0 | 1
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Ulcerative Keratitis (Eye disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The agreement is between the Sponsor and the sites, and restricts all use of trial related content and results for the duration of the trial until contractual obligations are superseded. The Sponsor has sole rights to all trial related content and results, and all PIs must gain permission to utilize the results.

DOCUMENTS (2):
  • Study Protocol (2021-05-04): https://cdn.clinicaltrials.gov/large-docs/46/NCT04485546/Prot_002.pdf
  • Statistical Analysis Plan (2021-05-20): https://cdn.clinicaltrials.gov/large-docs/46/NCT04485546/SAP_003.pdf